CLINICAL TRIAL: NCT06462001
Title: BCG + MMC: Adding Mitomycin C to BCG as Adjuvant Intravesical Therapy for High-risk, Non-muscle-invasive Bladder Cancer: a Randomised Phase 3 Trial
Brief Title: BCG + MMC: Adding Mitomycin C to BCG in High-risk, Non-muscle-invasive Bladder Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Collaborators: Australian and New Zealand Urogenital and Prostate Cancer Trials Group (Other); University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18UR004
Record Dates: First submitted 2023-12-29; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Transitional Cell Carcinoma; Transurethral Resection
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Mitomycin

STUDY DESIGN:
Intervention Model Description: an open label, randomised, stratified, 2-arm multicentre phase 3 clinical trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Standard Intravesical BCG (Active Comparator): Standard intravesical BCG therapy given as per usual standard of care
  Interventions: Biological: Bacillus Calmette-Guerin Vaccine Intravesical
- Arm B: Experimental BCG + MM (Experimental): Combination therapy with BCG and MM, given on specific protocol sessions
  Interventions: Biological: Bacillus Calmette-Guerin Vaccine Intravesical; Drug: Mitomycin

INTERVENTIONS:
Biological: Bacillus Calmette-Guerin Vaccine Intravesical — BCG (Oncotice) is administered intravesically as per usual standard of care
Drug: Mitomycin — MMC is administered intravesically as per usual standard of care
  Arms: Arm B: Experimental BCG + MM

SUMMARY:
Instillation of Bacillus of Calmette-Guerin (BCG) into the urinary bladder (intravesical administration) improves rates of disease recurrence and progression after transurethral resection (TUR) of high risk, non-muscle-invasive bladder cancer (NMIBC), but over 30% of people still develop recurrent transitional cell carcinoma (TCC) despite optimal therapy with adjuvant intravesical BCG. Our meta-analysis, including a recent randomised phase 2 trial, suggests that outcomes might be improved further by using an adjuvant intravesical regimen that includes both Mitomycin (MM) and BCG. These promising findings require corroboration in a definitive, large scale, randomised phase 3 trial using standard techniques for intravesical administration.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with confirmed high grade pTa or stage pT1 (any grade) non-muscle invasive bladder cancer on initial or re-resection histology (concurrent carcinoma in situ is allowed).
2. Age ≥ 18 yrs
3. No macroscopically visible disease at cystoscopy within 8 weeks prior to randomisation. This may either be the initial TURBT at which the primary tumour was completely resected, or a planned second cystoscopy and/ or re-resection done within 8 weeks of the initial TURBT.
4. ECOG Performance Status of 0-2
5. Adequate bone marrow, renal and liver function confirmed by pre-randomisation blood tests.
6. Study treatment both planned and able to start within 4 weeks of randomisation
7. Is willing to complete HRQL questionnaires or is unable to complete them because of literacy, insufficient English or limited vision
8. Willing and able to comply with all study requirements, including treatment, timing and/or nature of all required assessments
9. Signed, written informed consent

Exclusion Criteria:

1. Contraindications or hypersensitivity to investigational products, BCG and MM
2. Prior treatment with any other intravesical agent including BCG or MM (excludes single doses given post TURBT)
3. Current or past transitional cell carcinoma (TCC) of the upper urinary tract
4. Prior muscle-invasive (stage T2 or higher) transitional-cell carcinoma of the bladder
5. Bladder dysfunction precluding intravesical therapy e.g. Severe urinary incontinence or overactive or spastic bladder
6. Life expectancy < 3 months
7. Congenital or acquired immune deficiencies, whether due to a concurrent disease (e.g. acquired immune deficiency syndrome (AIDS), leukaemia, lymphoma) or immunosuppressive therapy (e.g. corticosteroids), or cancer therapy (cytotoxic drugs, radiation)
8. Prior radiotherapy of the pelvis
9. Prior or current treatment with radiotherapy-response or biological-response modifiers
10. Clinical evidence of existing active tuberculosis
11. History of another malignancy within 5 years prior to registration. Patients with non-melanomatous carcinoma of the skin are eligible for this study.
12. Serious medical or psychiatric conditions that might limit the ability of the patient to comply with the protocol.
13. Pregnancy, lactation, or inadequate contraception. Women must be post menopausal, infertile, or use a reliable means of contraception. Women of childbearing potential must have a negative pregnancy test done within 7 days prior to registration. Men must have been surgically sterilised or use a (double if required) barrier method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 5 years follow up
  Death, disease free survival, or evidence of transitional cell carcinoma (TCC)

SECONDARY OUTCOMES:
Activity | 3 months
  Clear cystoscopy at 3 months
Time to Recurrence | 5 years follow up
  Recurrence of TCC bladder
Time to Progression | 5 years follow up
  Recurrence of Higher Grade or Stage
Safety and adverse events | During treatment phase of the trial (typically 12 months)
  Adverse Events Graded According to CTC AE V4.03
Health-Related Quality of Life | 5 years follow up
  QLQ-BLS24. Individual internationally-validated (but subjective) symptom score questionnaire that gives an overall QOL assesment, that can be tracked throughout follow up. They do not use SI units of measurement.
Health-Related Quality of Life | 5 years follow up
  QLQ-C30. Individual internationally-validated (but subjective) symptom score questionnaire that gives an overall QOL assesment, that can be tracked throughout follow up. They do not use SI units of measurement.
Health-Related Quality of Life | 5 years follow up
  I-PSS. Individual internationally-validated (but subjective) symptom score questionnaire that gives an overall QOL assesment, that can be tracked throughout follow up. They do not use SI units of measurement.
Overall Survival Time | 5 years follow up
  Death from any Cause
Feasibility as a future standard of care | During treatment phase of the trial, typically 1 year
  Compliance with intravesical therapy, measured in percent (%) of planned intravesical therapies actually given
Marginal Resource Use | 5 years follow up
  Number of GP visits, Number of outpatient and emergency department visits, number of inpatient admissions and number of days admitted

OTHER OUTCOMES:
To consider future exploratory biomarker studies as potential prognostic biomarkers or predictive biomarkers of treatment | 5 years follow up
  Future (as yet unidentified) biomarker expression could be measured and then statistical association of those biomarkers with primary outcome meaures assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Dickon Hayne, PhD, Study Director — The University of Western Australia
Locations (1):
- Nottingham University Hospitals, Nottingham, United Kingdom